CLINICAL TRIAL: NCT00157768
Title: IRIS - Immediate Risk-stratification Improves Survival - Joint Study of the German University Hospitals and German Society of Leading Cardiological Hospital Physicians (ALKK)
Brief Title: IRIS : Use of Implantable Defibrillator in High-risk Patients Early After Acute Myocardial Infarction
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Collaborators: AstraZeneca (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: Medtronic_BRC_CRM_002
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2025-07-03 (Actual); Status verified 2018-10

CONDITIONS: Acute Myocardial Infarction
Keywords: Acute myocardial infarction; Non-sustained ventricular tachycardia; Left ventricular dysfunction; Implantable cardioverter defibrillator; ICD; Risk-stratification
MeSH Terms: conditions — Ventricular Dysfunction, Left | interventions — Defibrillators, Implantable

INTERVENTIONS:
Device: Implantable cardioverter defibrillator

SUMMARY:
Of the patients who survive hospitalization after an acute myocardial infarction, ca. 10% die of sudden cardiac death in the following 2 years. The prognosis appears not improved by medication with antiarrhythmics (class I/III). A positive effect of beta-blockers (Metoprolol CR/Zok) on total mortality after myocardial infarction in patients with heart failure is well established. On the other hand, an implantable defibrillator (ICD) proved to be superior to medication when used for secondary prevention in patients after cardiac arrest. The question arises whether ICD therapy is also effective in primary prevention in high risk patients after acute myocardial infarction. This study determines if patients, who were defined as high risk patients in the early post infarction phase by means of noninvasive methods, benefit from primary prevention by means of an ICD. Special emphasis is put on an individual optimization of the infarction therapy, including beta-blockers.

ELIGIBILITY:
Inclusion Criteria:

* acute myocardial infarction (5-31 days)
* fulfill requirement I and/or II :

  * I first ECG heart rate >= 90 bpm (within day 1-2 post MI) and LVEF <= 40 % (within day 5-31 post-MI)
  * II >= 1 episode of non-sustained ventricular tachycardia >= 150 bpm (on Holter, within 5-31 days post-MI)

Exclusion Criteria:

* Patients with ventricular arrhythmia, requiring clinical therapy, before the index infarction or more than 48 h later
* Patients with therapy refractory heart failure (NYHA IV)
* Myocardial infarction older than 31 days
* First-ECG not available or was recorded more than 48 h after the symptom onset.
* Patients with indication for CABG operation before inclusion
* Patients with cerebral organic psycho syndrome
* Secondary diseases which clearly limit life expectancy
* Patient with right sided artificial heart valve
* Patients with poor compliance
* Patients who are participating in another study
* Unstable clinical condition
* Pregnancy
* No consent from patient

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 900 (Estimated)
Dates: Start 1999-06-09 (Actual); Primary Completion 2007-10-15 (Actual); Study Completion 2007-10-15 (Actual)

PRIMARY OUTCOMES:
The null hypothesis is that all cause mortality in the treatment (Implantable cardioverter defibrillator =ICD) and control group is identical. The alternative hypothesis is that all cause mortality in the ICD group and control group is different.

SECONDARY OUTCOMES:
Type of death, Arrhythmic events, Serious cardiac and cerebral interventions,
Device-related complications, Hospitalizations, Quality of life

CONTACTS AND LOCATIONS:
Overall Officials: D. Andresen, Prof., Principal Investigator — Klinikum am Urban, Berlin, Germany; J. Senges, Prof., Principal Investigator — Herzzentrum Ludwigshafen, Germany; G. Steinbeck, Prof., Principal Investigator — Klinikum Grosshadern, Munich, Germany
Locations (1):
- Medtronic Bakken Research Center B.V., Maastricht, Netherlands

REFERENCES:
- [Derived] Steinbeck G, Andresen D, Seidl K, Brachmann J, Hoffmann E, Wojciechowski D, Kornacewicz-Jach Z, Sredniawa B, Lupkovics G, Hofgartner F, Lubinski A, Rosenqvist M, Habets A, Wegscheider K, Senges J; IRIS Investigators. Defibrillator implantation early after myocardial infarction. N Engl J Med. 2009 Oct 8;361(15):1427-36. doi: 10.1056/NEJMoa0901889. PMID 19812399